CLINICAL TRIAL: NCT06740877
Title: Relationship Between Skeletal Muscle Index in Preoperative Computed Tomography and a Neuromuscular Blocking Agent Dose Required for Maintaining Deep Neuromuscular Blockage: a Prospective Observational Study.
Brief Title: Skeletal Muscle Index and a Neuromuscular Blocking Agent
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Park InSun, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2501-947-303
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the recent development of image analysis, it has become possible to measure the skeletal muscle index representing the subject's muscle mass from preoperative computed tomography (CT) images. Therefore, in this study, the investigators quantify the skeletal muscle index from preoperative CT images and analyze the correlation with the dose of neuromuscular blocking agent, rocuronium, required for maintaining deep neuromuscular blockade.

DETAILED DESCRIPTION:
Deep neuromuscular blockade improves the condition of surgeon's surgical field during the surgery and reduces the acute postoperative pain. The dosage of neuromuscular blocking agent has been usually administered according to the patient's actual body weight, but even with the same body weight, the ratio of muscle to fat varies from individual to individual, and there are many differences depending on age, gender, and exercise level.

Therefore, if the dose of neuromuscular blocking agent is administered according to actual body weight, additional doses may be required due to insufficient neuromuscular blockade, or excessive doses may occur. However, it was difficult to quantify the muscle mass, with the recent development of image analysis, it has become possible to measure the skeletal muscle index representing the subject's muscle mass from preoperative computed tomography (CT) images. Therefore, in this study, the investigators quantify the skeletal muscle index from preoperative CT images and analyze the correlation with the dose of neuromuscular blocking agent, rocuronium, required for maintaining deep neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily agreed and signed the written consent form before participating in the study
* American Society of Anesthesiologists physical class (ASA class) 1-3
* Patients scheduled for elective colon surgery under general anesthesia
* Patients undergoing abdominal computed tomography for routine preoperative preparation

Exclusion Criteria:

* Pregnant women
* Decreased renal function (GFR<60mL/min/1.73m2).
* Patients taking drugs that affect deep neuromuscular blockade
* Patients with a history of neuromuscular and muscle disorders

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective colon surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle index | preoperative period
  Muscle amount

CONTACTS AND LOCATIONS:
Overall Officials: Insun Park, M.D./Ph.D., Principal Investigator — assistant professor